CLINICAL TRIAL: NCT07286461
Title: VIROMARKERS GA n.101194735 - CMV and TTV Biomarkers Study Protocol
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: Heinrich-Heine-Universitaet Duesseldorf (Unknown)
Responsible Party: Principal Investigator, Valentina Svicher, Professor, University of Rome Tor Vergata
Other Study IDs: 101194735-CMV-TTV
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient; CMV
Keywords: CMV; TTV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A blood sample will be obtained for all participants at enrollment to be shipped to a central repository for testing.
  In all samples resulting positive to CMV-DNAemia, an additional aliquot of the same sample will be pre-treated with DNase prior to DNA extraction, to exclude DNA which is not protected by a viral capsid (e.g., concatemeric DNA) from Real Time-PCR amplification, thus inducing the loss of non-infectious viral DNA.
  The quantification of CMV-RNA and TTV-DNAemia will be carried at T0 and every month during and after letermovir prophylaxis up to the end of study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- receiving HSCT and being seropositive for CMV, receiving HSCT from a donor CMV positive: The sibjects going to be enrolled are:
  Having received or due to receive HSCT; HSCT recipient is seropositive for CMV, or receiving HSCT from a CMV seropositive donor
  Interventions: Drug: letermovir prophylaxis

INTERVENTIONS:
Drug: letermovir prophylaxis — quantification of CMV-DNA in blood or plasma by using Real-Time PCR assays

SUMMARY:
The study is one of the researches carried out in the VIROMARKERS Project.

The project VIROMARKERS is supported by the Innovative Health Initiative Joint Undertaking (IHI JU) under grant agreement No 101194735. The JU receives support from the European Union's Horizon Europe research and innovation programme and COCIR, EFPIA, Europa Bio, MedTech Europe, Vaccines Europe, and Roboscreen.

To date, the virological surveillance for CMV replication relies basically on the quantification of CMV-DNA in blood or plasma by using Real-Time PCR assays, and CMV-DNAemia is known to correlate with both CMV-related disease and non-relapse mortality [Ljungman, 2025]. However, the detection of CMV-DNAemia is not always associated with an active CMV replication, particularly in patients exposed to letermovir. Therefore, the identification of new virological markers to accurately monitor CMV activity in the early and late post-HSCT phases, remains a crucial issue especially in individuals receiving letermovir as prophylaxis to ensure a proper diagnosis of CMV infection/disease and to guide prophylactic and pre-emptive antiviral treatment.

In this setting, the quantification of CMV-RNA represents a potential candidate marker capable of better reflecting the presence of complete, infectious CMV virions than CMV-DNAemia. Despite several data support a correlation of CMV UL21.5-mRNA with viral activity [Nicastro, 2025], studies investigating the kinetics of this viral mRNA among immune-suppressed patients at risk of CMV re-uptake are largely missing, especially in the setting of patients receiving antiviral prophylaxis with letermovir after HSCT.

TTV-DNA load was mostly investigated in solid organ transplant patients (SOT), where it showed a good correlation of high viral load and degree of immunosuppression. In HSCT patients the interaction of the immune system, which is under reconstitution, and clinically relevant CMV infection is more complex. First data have been reported by our group [Gilles et al., 2017] showing high TTV load as a prognostic marker for risk of complications after HSCT. Little information is available for HSCT patients under letermovir prophylaxis.

Specific primary objectives related to CMV monitoring in the HSCT setting are the following:

Primary In participants who received HSCT, to estimate the rate of initiation of anti-CMV therapy during letermovir-based prophylaxis and the rate of CMV re-activation (based on symptoms, signs of organ dysfunction and CMV-DNAemia) after suspension of letermovir.

To evaluate the kinetics of CMV-RNAemia, CMV-DNAemia and TTV-DNAemia and their correlation during prophylaxis with letermovir.

To establish whether early quantitative CMV-RNA level or the early kinetics of CMV-RNAemia and TTV-DNAemia during prophylaxis can predict initiation of anti-CMV therapy.

In participants not initiating anti-CMV therapy during prophylaxis, to establish whether quantitative CMV-RNA level at time of letermovir suspension or the kinetics of CMV-RNAemia and TTV-DNAemia during prophylaxis can predict CMV re-activation (based on symptoms signs of organ dysfunction and CMV-DNAemia) after suspension of letermovir.

Secondary objectives include to establish a cut-off for CMV-RNAemia and TTV DNAemia to maximize the accuracy of prediction of CMV re-activation after suspension of prophylaxis; to explore the kinetics of CMV-RNAemia and TTV-DNAemia in participants treated with anti CMV drugs.

The information used from this study on participants in the HSCT setting will be rapidly analyzed and shared broadly to guide policymakers for the use and monitoring of CMV-DNAemia, CMV-RNAemia and TTV-DNAemia in CMV disease and to design future studies. For exact plans regarding the expected date of study completion and plans for dissemination please refer to separate documents produced within the WP5 of VIROMARKERS.

DETAILED DESCRIPTION:
Human cytomegalovirus (CMV) infection represents a major cause of morbidity and mortality after allogeneic hematopoietic stem cell transplantation (HSCT), mainly occurring as viral reactivation from latency in seropositive patients but also as de novo infection in HSCT recipients from seropositive donors. Indeed, CMV infection is a frequent event following HSCT and can cause severe end-organ disease (pneumonia, colitis, retinitis, hepatitis), as well as an increased risk of graft versus host disease (GVHD) and bacterial/fungal superinfections, overall responsible for a high transplant-related morbidity and mortality [Ljungman, 2025].

Recently, anti-CMV prophylaxis has substantially reduced the risk of CMV infection and disease, as well as its related mortality [Einsele, 2020]. To date, anti-CMV prophylaxis is mainly based on the usage of letermovir, an inhibitor of CMV terminase complex, that selectively blocks the cleavage of the concatemeric progeny CMV-DNA to single mature CMV genomes and is then associated with a limited drug toxicity [Ljungman, 2025]. Although letermovir prophylaxis has been demonstrated to be safe and effective at reducing CMV disease and mortality at early times post-HSCT, late CMV infection occurring after prophylaxis suspension (upon 100 days post-HSCT) continues to represent a major concern for patients undergoing HSCT [Ljungman, 2025].

Participant Selection

To be eligible for enrollment participants must be ≥ 18 years of age, have a signed informed consent, and fulfill all of the following criteria:

Having received or due to receive HSCT HSCT recipient is seropositive for CMV, or receiving HSCT from a CMV seropositive donor Eligible to receive antiviral prophylaxis with letermovir for preventing CMV infection for at least 100 days in Italy or 200 days in Germany after HSCT according to the current guidelines.

Study Plan Participants will be enrolled at participating clinical sites. At the time of receiving HSCT (enrollment T0), demographics, medical history, medications and treatments prescribed will be recorded.

Participants will be monitored post HCST by clinical visits as well as laboratory tests using stored plasma samples. The collection of samples will be based according to the duration of letermovir prophylaxis which varies by country: 100 days in Italy vs. 200 days in Germany. See Appendix B for the time schedule of plasma samples collection according to country of enrolment.

In all samples resulting positive to CMV-DNAemia, an additional aliquot of the same sample will be pre-treated with DNase prior to DNA extraction, to exclude DNA which is not protected by a viral capsid (e.g., concatemeric DNA) from Real Time-PCR amplification, thus inducing the loss of non-infectious viral DNA. The quantification of TTV-DNAemia will be carried at T0 and every month during and after letermovir prophylaxis up to the end of study period.

Proposed research utilizing stored clinical specimens collected per this protocol will be reviewed and approved by the Protocol Team, the VIROMARKERS Scientific Steering Committee, and EC Horizon Europe.

Background and Rationale Human cytomegalovirus (CMV) infection represents a major cause of morbidity and mortality after allogeneic hematopoietic stem cell transplantation (HSCT), mainly occurring as viral reactivation from latency in seropositive patients but also as de novo infection in HSCT recipients from seropositive donors. Indeed, CMV infection is a frequent event following HSCT and can cause severe end-organ disease (pneumonia, colitis, retinitis, hepatitis), as well as an increased risk of graft versus host disease (GVHD) and bacterial/fungal superinfections, overall responsible for a high transplant-related morbidity and mortality.

In the setting of HSCT, CMV infection develops in >60% of CMV seropositive recipients (R+), and in approximately 10% of seronegative recipients (R-) transplanted from seropositive donors (D+) [George et al., 2010], in absence of any preventive strategy. Recently, anti-CMV prophylaxis has substantially reduced the risk of CMV infection and disease, as well as its related mortality [Einsele, 2020]. To date, anti-CMV prophylaxis is mainly based on the usage of letermovir, an inhibitor of CMV terminase complex, that selectively blocks the cleavage of the concatemeric progeny CMV-DNA to single mature CMV genomes and is then associated with a limited drug toxicity [Deleenheer, 2018]. Although letermovir prophylaxis has been demonstrated to be safe and effective at reducing CMV disease and mortality at early times post-HSCT, late CMV infection occurring after prophylaxis suspension (upon 100 days post-HSCT) continues to represent a major concern for patients undergoing HSCT.

Recently EMA and FDA approved letermovir prophylaxis for 200 days instead of 100, which further decreases the risk of clinically relevant CMV infection (PREVYMIS, INN-letermovir). Nevertheless, the availability of accurate virological markers to accurately monitor CMV activity in the early and late post-HSCT phases, remains a crucial issue to ensure a proper diagnosis of CMV infection and disease and to guide prophylactic and pre-emptive antiviral treatment.

With this regard, to date, the virological surveillance for CMV replication relies basically on the quantification of CMV-DNA in blood or plasma by using Real-Time PCR assays [Ljungman, 2025], and CMV-DNAemia is known to correlate with both CMV-related disease [Ljungman, 2025] and non-relapse mortality.

However, the detection of CMV-DNAemia is not always associated with an active CMV replication, particularly in patients exposed to letermovir as prophylaxis since this drug, acting as an inhibitor of viral terminase, does not inhibit viral DNA synthesis but only its further maturation into individual genomes. In particular, a recent study from Baldanti's group, demonstrated that CMV DNAemia during LMV prophylaxis can be positive even in absence of complete CMV replicative cycles, since non-infectious CMV-DNA are released from degrading abortively infected cells even in the absence of infectious virions. This issue is particularly relevant since the interpretation of CMV-DNAemia as active viral replication can lead to a potential overestimation of CMV infection during prophylaxis and to a consequent unjustified switch to high-toxicity antivirals as ganciclovir in a high proportion of patients.

Thus, the implementation of CMV diagnostics with the use of novel markers, capable of reflecting more accurately CMV replicative activity, represents a still unmet need that can significantly improve the management of CMV risk in patients undergoing HSCT.

In this setting, the quantification of CMV-RNA represents a potential candidate marker capable of better reflecting the presence of complete, infectious CMV virions.

In particular, the currently available assay for CMV-RNA quantification (EliTech) targets the UL21.5 spliced CMV mRNA, a late viral mRNA that has been demonstrated to be packaged within the circulating complete CMV virions [Nicastro, 2025]. Despite several data support a correlation of CMV UL21.5-mRNA with viral activity, studies investigating the kinetics of this viral mRNA among immune-suppressed patients at risk of CMV re-uptake are largely missing, even more in the setting of patients receiving antiviral prophylaxis with letermovir after HSCT.

Methodology Study Design This observational study will include at least 290 consecutive patients undergoing HSCT at risk of CMV infection. Clinical management of participants will be carried out according to international and local guidelines, without any modification due to the current study. Participants will be followed for the entire duration of prophylaxis treatment followed by a minimum of 3 months after suspension.

Endpoint definitions

Before suspension of prophylaxis with letermovir:

Clinically significant CMV infection requiring initiation of anti-CMV drugs: defined as CMV end-organ disease or any CMV-related clinical event, based on CMV-DNAemia (>1,000 IU/ml is the cut-off generally used by haematologists in Italy) and the clinical condition of the patient. These include the following clinical symptoms: neurological, gastrointestinal, pneumonia, retinitis.

After suspension of prophylaxis with letermovir (relapses):

CMV infection: defined as CMV-DNAemia >112IU/ml (lower limit of quantification [LLOQ] by the commercially available Real-Time EliTech CMV DNA ELITe MGB® Kit assay used at UTOV) in seropositive HSCT recipients and in seronegative Participants receiving HSCT from seropositive donors according to the criteria recommended by the CMV Drug Development Forum.

Clinically significant CMV infection: defined as CMV end-organ disease or any CMV-related clinical symptoms (neurological, gastrointestinal, pneumonia, retinitis, see above), based on documented DNAemia >112 IU/ml and the clinical condition of the patient.

a single value of CMV-DNAemia >1,000 IU/ml or with CMV-DNAemia increasing from 500 to 1,000 IU/ml without symptoms of CMV-related disease Participants with any CMV-DNAemia with symptoms of CMV-related disease will start a therapy based on gancyclovir, valganciclovir and other second line treatments (such as foscarnet, maribavir or letermovir-gancyclovir combination) for CMV-disease, according to the virological and clinical response. Dosage will be assessed based on renal function in terms of creatinine clearance. In cases of persistent or growing values of CMV viremia under ganciclovir treatment (suspected for clinical resistance) the switch to other antivirals (i.e. Foscarnet) will be evaluated, according to current guidelines.

Study Objectives Primary and secondary objectives are stated below. Primary In participants who received HSCT, to estimate the rate of initiation of anti-CMV therapy during letermovir-based prophylaxis and the rate of CMV reactivation (based on symptoms, signs of organ dysfunction and CMV-DNAemia) after suspension of letermovir.

To evaluate the kinetics of CMV-RNA, CMV-DNAemia and TTV-DNAemia and their correlation during prophylaxis with letermovir.

To establish whether early quantitative CMV-RNA level or the early kinetics of CMV-RNA and TTV-DNAemia during prophylaxis can predict initiation of anti-CMV therapy.

In participants not initiating anti-CMV therapy during prophylaxis, to establish whether quantitative CMV-RNA level at time of letermovir suspension or the kinetics of CMV-RNA and TTV-DNAemia during prophylaxis can predict CMV re-activation (based on symptoms signs of organ dysfunction and CMV-DNAemia) after suspension of letermovir.

Secondary To establish a cut-off for CMV-RNA levels and TTV DNAemia To maximize the accuracy of prediction of CMV re-activation after suspension of prophylaxis.

To explore the kinetics of CMV-RNAemia and TTV-DNAemia in participants treated with anti CMV drugs.

To explore the correlation between CMV-RNAemia and CMV-DNAemia after considering concatemeric DNA estimated from pre-treating the sample with DNase prior to DNA extraction Data collected to address these objectives will be rapidly analyzed and summarized so that more targeted protocols for treatment and monitoring of the response can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Be > 18 years of age
* Sign an informed consent
* HSCT recipients seropositive to CMV, or receiving HSCs from a CMV seropositive donor
* Antiviral prophylaxis with letermovir for preventing CMV infection will be administered for 100 days in Italy (or 200 days in Germany) after HSCT to all participants according to the current guidelines

Exclusion Criteria:

Individuals <18 years old undergoing HSCT Individuals not receiving letermovir prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will include at least 290 consecutive patients undergoing HSCT at risk of CMV infection. Clinical management of participants will be carried out according to international and local guidelines, without any modification due to the current study. Participants will be followed for the entire duration of prophylaxis treatment followed by a minimum of 3 months after suspension.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
CMV-DNA | Italy: 0 , 7, 15, 30, 45, 60, 75, 90,100 107 115,130, 145, 160, 175, 190 day post HSCT). Germany:0, 7, 15, 30, 60, 90, 120, 150, 180 , 200 , 207 230, 260, 290 day post HSCT
  plasma samples will be collected at the following time-points for CMV-RNA quantification

CONTACTS AND LOCATIONS:
Overall Officials: VALENTINA SVICHER, Study Chair — UNIVERST' DI ROMA TOR VERGATA
Locations (1):
- Heinrich-Heine-Universitaet Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Yes
The access to the data, both for view, upload and download will be monitored with "Access control logging", based on a user authentication control with geolocalization of the access, based, for example, on Google authenticated accounts - Google Workspace or similar.
  The repository of the database will be located on the INFORMAPRO/EURESIST organization Google WorkSpace Shared Drive infrastructure, located in the EU space, as the organizations are Italian and by contract, the hosted workspace is inside the EU space.
  In order to make the data interoperable, it is important to have 3 basic features:
  A STANDARDIZED Metadata. This standardization has to be developed with the common efforts of all WP participated partners

REFERENCES:
- [Background] Gilles R, Herling M, Holtick U, Heger E, Awerkiew S, Fish I, Holler K, Sierra S, Knops E, Kaiser R, Scheid C, Di Cristanziano V. Dynamics of Torque Teno virus viremia could predict risk of complications after allogeneic hematopoietic stem cell transplantation. Med Microbiol Immunol. 2017 Oct;206(5):355-362. doi: 10.1007/s00430-017-0511-4. Epub 2017 Jul 12. PMID 28702856
- [Background] Nicastro E, Severi E, Passera I, Totaro M, Matarazzo L, Fornataro L, Morotti F, Tebaldi A, Bonanomi E, Bravi M, Di Giorgio A, Covini S, Dolci M, Pinelli D, Arosio MEG, D'Antiga L. Cytomegalovirus-RNA Accurately Identifies Clinically Significant Infection Needing Preemptive Therapy in Liver Transplanted Children: A Proof-of-Concept Study. J Med Virol. 2025 Apr;97(4):e70347. doi: 10.1002/jmv.70347. PMID 40232168
- [Background] Cassaniti I, Colombo AA, Bernasconi P, Malagola M, Russo D, Iori AP, Girmenia C, Greco R, Peccatori J, Ciceri F, Bonifazi F, Percivalle E, Campanini G, Piccirilli G, Lazzarotto T, Baldanti F. Positive HCMV DNAemia in stem cell recipients undergoing letermovir prophylaxis is expression of abortive infection. Am J Transplant. 2021 Apr;21(4):1622-1628. doi: 10.1111/ajt.16450. Epub 2021 Feb 8. PMID 33320429
- [Background] Ljungman P, Alain S, Chemaly RF, Einsele H, Galaverna F, Hirsch HH, Sadowska-Klasa A, Navarro D, Styczynski J, de la Camara R. Recommendations from the 10th European Conference on Infections in Leukaemia for the management of cytomegalovirus in patients after allogeneic haematopoietic cell transplantation and other T-cell-engaging therapies. Lancet Infect Dis. 2025 Aug;25(8):e451-e462. doi: 10.1016/S1473-3099(25)00069-6. Epub 2025 Apr 3. PMID 40188837